CLINICAL TRIAL: NCT01776840
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor, PCI-32765 (Ibrutinib), in Combination With Bendamustine and Rituximab (BR) in Subjects With Newly Diagnosed Mantle Cell Lymphoma
Brief Title: A Study of the Bruton's Tyrosine Kinase Inhibitor Ibrutinib Given in Combination With Bendamustine and Rituximab in Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100967; PCI-32765MCL3002 (Other: Janssen Research & Development, LLC); U1111-1137-0389 (Other: Universal Trial Number); 2012-004056-11 (EudraCT Number)
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2022-07-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Ibrutinib; Bruton's tyrosine kinase inhibitor; Bendamustine hydrochloride; Rituximab
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; Rituximab; ibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Placebo Comparator)
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Placebo
- Treatment Arm B (Experimental)
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Bendamustine — 90 mg/m2 administered intravenously on Days 1-2, Cycles 1-6
Drug: Rituximab — 375 mg/m2 administered intravenously on Day 1, Cycles 1-6; if complete response or partial response is achieved, 375 mg/m2 is administered on Day 1 of every second cycle for a maximum of 12 additional doses
Drug: Ibrutinib — 560 mg (4 x 140 mg capsules) administered orally once daily continuously starting on Day 1, Cycle 1 until disease progression, or unacceptable toxicity, or study end
  Arms: Treatment Arm B
Drug: Placebo — 4 capsules administered orally once daily continuously starting on Day 1, Cycle 1 until disease progression, or unacceptable toxicity, or the final analysis of progression-free survival
  Arms: Treatment Arm A

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ibrutinib given in combination with bendamustine and rituximab in patients 65 years of age or older with newly diagnosed mantle cell lymphoma.

DETAILED DESCRIPTION:
This is a randomized (individuals assigned to study treatment by chance), double blind (neither physician nor participant knows the treatment that the participant receives), placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial)-controlled study to compare the efficacy and safety of ibrutinib given in combination with bendamustine and rituximab (BR) with BR alone in participants newly diagnosed with mantle cell lymphoma (MCL) who are 65 years of age or older. Approximately 520 participants will be randomly assigned in a 1:1 ratio and stratified by simplified Mantle Cell Lymphoma International Prognostic Index (MIPI) score (low risk [0-3] versus intermediate risk [4-5] versus high risk [6-11]). The treatment phase will extend from randomization until discontinuation of all study treatment or the clinical cutoff for the end of study. A cycle is defined as 28 days. All participants will receive open-label (identity of assigned study drug will be known) BR background therapy for a maximum of 6 cycles; participants with a complete response or partial response will continue to receive open-label background therapy with rituximab maintenance every second cycle for a maximum of 12 additional doses. In addition to the background therapy, all participants will receive blinded study drug (ibrutinib or placebo). Participants randomized to treatment Arm A will receive placebo capsules and participants randomized to treatment Arm B will receive ibrutinib capsules. Study drug will be administered daily and continuously until disease progression, unacceptable toxicity, or study end. Participants with stable disease after initial chemoimmunotherapy (BR+ibrutinib/placebo) should continue treatment with ibrutinib/placebo until disease progression, unacceptable toxicity, or study end. Participants with progressive disease must discontinue all study treatment. For participants who discontinue background therapy and do not have progressive disease, treatment with study drug will continue until disease progression or unacceptable toxicity or the clinical cutoff for the final analysis of progression-free survival (PFS). Participants receiving BR, rituximab, or ibrutinib at the clinical cutoff for the final analysis of PFS will continue open-label treatment until disease progression or unacceptable toxicity. Placebo will be stopped when the study is unblinded for the clinical cutoff for the final analysis of PFS. The posttreatment follow-up phase will begin once a participant discontinues bendamustine and rituximab and study drug. Participants who discontinue for reasons other than disease progression must continue to have disease evaluations as outlined in the protocol. Participants who discontinue due to disease progression will be followed for survival and subsequent anti-MCL therapy. The posttreatment follow-up phase will continue until death, lost to follow up, consent withdrawal, or study end, whichever occurs first. Four clinical cutoffs are planned. The first 3 clinical cutoffs will occur when approximately 134, 180, and 265 PFS events have been observed, respectively. The interim analyses and the final analysis of PFS will take place at these 3 clinical cutoffs, respectively; participant treatment assignment will be unblinded and placebo treatment will be stopped at the clinical cutoff for the final analysis of PFS. Treatment unblinding and stopping of placebo treatment could occur before the planned final analysis of PFS if recommended by the independent Data Monitoring Committee (DMC) after an interim analysis. The last cutoff will occur at the end of study, when 60% of the randomized participants have died or the Sponsor terminates the study, whichever comes first. Efficacy assessments will be conducted in accordance with the Revised Response Criteria for Malignant Lymphoma. Safety will be monitored throughout the study and summarized. Blood samples will be drawn for assessment of pharmacokinetic parameters. Blood and bone marrow will be collected for assessment of minimal residual disease and biomarker studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mantle cell lymphoma (MCL) reviewed and approved by central laboratory: diagnosis must include morphology and expression of either cyclin D1 in association with other relevant markers (eg, CD19, CD20, PAX5 and CD5) or evidence of t(11;14) as assessed by cytogenetics, fluorescent in situ hybridization (FISH), or polymerase chain reaction (PCR)
* Clinical Stage II, III, or IV by Ann Arbor Classification
* At least 1 measurable site of disease according to Revised Response Criteria for Malignant Lymphoma
* No prior therapies for MCL
* Eastern Cooperative Oncology Group (ECOG) performance status grade 0 or 1
* Hematology and biochemical laboratory values within protocol-defined limits
* Agrees to protocol-defined use of effective contraception
* Negative blood or urine pregnancy test at screening

Exclusion Criteria:

* Major surgery within 4 weeks of random assignment
* Known central nervous system lymphoma
* Diagnosed or treated for malignancy other than MCL, except: malignancy treated with curative intent and with no known active disease present for >=3 years before random assignment; adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; adequately treated cervical carcinoma in situ without evidence of disease
* Patients for whom the goal of therapy is tumor debulking prior to stem cell transplant
* History of stroke or intracranial hemorrhage within 6 months prior to random assignment
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with strong CYP3A inhibitors
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Vaccinated with live, attenuated vaccines within 4 weeks of random assignment
* Known history of human immunodeficiency virus (HIV) or active hepatitis C virus or active hepatitis B virus infection or any uncontrolled active systemic infection requiring intravenous antibiotics
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 523 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (201):
- United States (44):
  - Tucson, Arizona
  - Burbank, California
  - La Jolla, California
  - Stanford, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Stamford, Connecticut
  - Chicago, Illinois
  - Maywood, Illinois
  - Niles, Illinois
  - Springfield, Illinois
  - Goshen, Indiana
  - Iowa City, Iowa
  - Sioux City, Iowa
  - Topeka, Kansas
  - Westwood, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Jefferson City, Missouri
  - Lincoln, Nebraska
  - Hackensack, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Hawthorne, New York
  - New York, New York
  - Durham, North Carolina
  - Greenville, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Eugene, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Watertown, South Dakota
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Burlington, Vermont
  - Spokane, Washington
  - Vancouver, Washington
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - La Capital
  - Paraná
- Australia (8):
  - Adelaide
  - Auchenflower
  - Box Hill
  - Concord
  - Douglas
  - Gosford
  - Hobart
  - Prahran
- Belgium (7):
  - Antwerp
  - Bruges
  - Brussels
  - Ghent
  - Leuven
  - Wilrijk
  - Yvoir
- Brazil (6):
  - Barretos
  - Goiânia
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - São Paulo
- Canada (5):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec
- China (6):
  - Beijing
  - Chengdu
  - Guangzhou
  - Hangzhou
  - Shanghai
  - Tianjin
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- France (7):
  - Créteil
  - F-75 730 Paris Cedex 15
  - Grenoble
  - Nantes
  - Paris
  - Pessac
  - Tours
- Germany (8):
  - Berlin
  - Heidelberg
  - Jena
  - Mainz
  - München
  - TÿBINGEN
  - Ulm
  - Villingen-Schwenningen
- Greece (3):
  - Athens
  - Athens Attica
  - Thessalonikis
- Hungary (5):
  - Budapest
  - Debrecen
  - Kaposvár
  - Pécs
  - Szeged
- Ireland (2):
  - Dublin
  - Galway
- Israel (9):
  - Afula
  - Beersheba
  - Haifa
  - Jerusalem
  - Nahariya
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
  - Ẕerifin
- Japan (9):
  - Fukuoka
  - Hiroshima
  - Kyoto
  - Nagoya
  - Osaka
  - Sapporo
  - Sendai
  - Suita
  - Tokyo
- Mexico (2):
  - Monterrey
  - Oaxaca City
- Netherlands (6):
  - Amsterdam-Zuidoost
  - Dordrecht
  - Groningen
  - Leiden
  - Rotterdam
  - Utrecht
- Poland (5):
  - Bydgoszcz
  - Krakow
  - Olsztyn
  - Warsaw
  - Wroclaw
- San Juan, Puerto Rico
- Russia (14):
  - Chelyabinsk
  - Krasnodar
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Petrozavodsk
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Sochi
  - St.Petersurg
  - Syktyvkar
  - Volgograd
  - Yekaterinburg
- Slovakia (5):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Martin
  - Prešov
- South Korea (3):
  - Gyeonggi-do
  - Jeollanam-do
  - Seoul
- Spain (6):
  - Barcelona
  - Madrid
  - Oviedo
  - Palma de Mallorca
  - Salamanca
  - Santiago de Compostela
- Sweden (5):
  - Linköping
  - Lund
  - Stockholm
  - Umeaa
  - Uppsala
- Taiwan (6):
  - Changhua
  - Kaohsiung County
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (7):
  - Adana
  - Ankara
  - Diyarbakır
  - Istanbul
  - Izmir
  - Kayseri
  - Mersin
- Ukraine (5):
  - Cherkassy
  - Donetsk
  - Khmelnitskiy
  - Kiev
  - Lviv
- United Kingdom (10):
  - Canterbury
  - Glasgow
  - Leeds
  - Leicester
  - Liverpool
  - London
  - Manchester
  - Plymouth
  - Southampton
  - Sutton

REFERENCES:
- [Derived] Wang ML, Jurczak W, Jerkeman M, Trotman J, Zinzani PL, Belada D, Boccomini C, Flinn IW, Giri P, Goy A, Hamlin PA, Hermine O, Hernandez-Rivas JA, Hong X, Kim SJ, Lewis D, Mishima Y, Ozcan M, Perini GF, Pocock C, Song Y, Spurgeon SE, Storring JM, Walewski J, Zhu J, Qin R, Henninger T, Deshpande S, Howes A, Le Gouill S, Dreyling M; SHINE Investigators. Ibrutinib plus Bendamustine and Rituximab in Untreated Mantle-Cell Lymphoma. N Engl J Med. 2022 Jun 30;386(26):2482-2494. doi: 10.1056/NEJMoa2201817. Epub 2022 Jun 3. PMID 35657079

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 523 subjects were randomized in this study.
Groups:
- Placebo + Bendamustine and Rituximab (BR) (Treatment A): Participants received 4 capsules of ibrutinib-matching Placebo administered orally once daily continuously starting on Day 1, Cycle 1 until disease progression, or unacceptable toxicity, or study end, whichever occurred first. All participants also received a maximum of 6 cycles of BR background therapy (bendamustine hydrochloride 90 milligrams per meter square [mg/m^2] intravenous [IV] infusion on Days 1 and 2 of each cycle and rituximab 375 mg/m^2 IV infusion on Day 1 of each cycle), unless disease progression or unacceptable toxicity prior to Cycle 6. Participants with a complete response (CR) or partial response (PR) continued to receive background therapy with rituximab maintenance (375 mg/m^2 IV infusion) on Day 1 every second cycle starting at Cycle 8 for a maximum of 12 additional doses unless disease progression or unacceptable toxicity. Each cycle was of 28 days. Participants received treatment A up to 100.1 months. After treatment unblinding at the time of the primary analysis, participants randomized to Treatment A discontinued placebo treatment.
- Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B): Participants received ibrutinib capsules 560 mg (4*140 mg capsule) administered orally once daily continuously starting on Day 1, Cycle 1 until disease progression, or unacceptable toxicity, or study end, whichever occurred first. All participants also received a maximum of 6 cycles of BR background therapy (bendamustine hydrochloride 90 mg/m^2 IV infusion on Days 1 and 2 of each cycle and rituximab 375 mg/m^2 IV infusion on Day 1 of each cycle), unless disease progression or unacceptable toxicity prior to Cycle 6. Participants with a CR or PR continued to receive background therapy with rituximab maintenance (375 mg/m^2 IV infusion) on Day 1 every second cycle starting at Cycle 8 for a maximum of 12 additional doses unless disease progression or unacceptable toxicity. Each cycle was of 28 days. Participants received treatment B up to 117.2 months. After treatment unblinding at the time of the primary analysis, participants randomized to Treatment B continued treatment with ibrutinib at the discretion of the investigator.
Period: Overall Study
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Started | 262 | 261
Safety Analysis Set (Treated) | 260 | 259
Completed (Participants who died were considered to have completed the study.) | 129 | 119
Not Completed | 133 | 142
Not completed — Lost to Follow-up | 12 | 7
Not completed — Withdrawal by Subject | 32 | 48
Not completed — Sponsor decision | 89 | 87

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B) | Total
Number analyzed (Participants) | 262 | 261 | 523
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (5.2) | 71.8 (5.04) | 71.7 (5.12)
Age, Customized [Count of Participants; unit: Participants]
  70 years and over | 154 | 162 | 316
  < 70 years | 108 | 99 | 207
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 83 | 159
  Male | 186 | 178 | 364
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 18 | 35
  Not Hispanic or Latino | 234 | 232 | 466
  Unknown or Not Reported | 11 | 11 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 42 | 47 | 89
  Black or African American | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 206 | 199 | 405
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 9 | 10 | 19
  Other | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 0 | 4 | 4
  AUSTRALIA | 12 | 19 | 31
  BELGIUM | 10 | 5 | 15
  BRAZIL | 10 | 11 | 21
  CANADA | 7 | 4 | 11
  CHINA | 26 | 31 | 57
  CZECH REPUBLIC | 8 | 7 | 15
  FRANCE | 13 | 8 | 21
  GERMANY | 5 | 3 | 8
  GREECE | 3 | 4 | 7
  HUNGARY | 5 | 5 | 10
  IRELAND | 0 | 2 | 2
  ISRAEL | 9 | 5 | 14
  ITALY | 13 | 13 | 26
  JAPAN | 4 | 7 | 11
  MEXICO | 2 | 1 | 3
  NETHERLANDS | 3 | 5 | 8
  POLAND | 17 | 18 | 35
  RUSSIAN FEDERATION | 12 | 15 | 27
  SLOVAKIA | 2 | 1 | 3
  SOUTH KOREA | 6 | 6 | 12
  SPAIN | 7 | 13 | 20
  SWEDEN | 9 | 9 | 18
  TAIWAN | 4 | 2 | 6
  TURKEY | 6 | 8 | 14
  UKRAINE | 5 | 6 | 11
  UNITED KINGDOM | 16 | 14 | 30
  UNITED STATES | 48 | 35 | 83

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the interval between the date of randomization to the date of disease progression (PD) or relapse from complete response (CR) or death, whichever was first reported. Disease assessments were based on the 2007 Revised Response Criteria for Malignant Lymphoma. PD was defined as any new lesion or increase by 50 percent (%) of previously involved sites from nadir (PD criteria: Appearance of new nodal lesion 1.5 centimeters [cm] in any axis, 50% increase in sum of product of diameters [SPD] of greater than [>] 1 node or 50% increase in longest diameter of previously identified node 1 cm in short axis).
Time Frame: Up to 97 months
Population: Intent-to-treat (ITT) analysis set included all randomized participants and classified according to the assigned treatment group, regardless of the actual treatment received. Here, N (overall number of participants analyzed) signifies number of participants that were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 262 | 261
months | 52.9 [43.7 to 71.0] | 80.6 [61.9 to NA] — Here, 'NA' refers that the upper limit of 95% confidence interval was not estimable because of small number of events.
Statistical Analysis 1: Comparison: Placebo + Bendamustine and Rituximab (BR) (Treatment A) vs Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B); Test type: Superiority; p = 0.011, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.59 to 0.96]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of the participant's death. Kaplan-Meier estimate was used.
Time Frame: From randomization (Day -3) up to 121 months
Population: ITT analysis set included all randomized participants and classified according to the assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 262 | 261
months | 95.9 [86.1 to 115.3] | 104.3 [81.1 to NA] — Here, 'NA' refers that the upper limit of 95% confidence interval was not estimable because of small number of participants with events.

3. Secondary Outcome: Complete Response Rate
Description: Complete response (CR) rate was defined as the percentage of participants who achieve CR (based on investigator assessment) on or prior to the initiation of subsequent anticancer therapy. Criteria for CR: disappearance of all evidence of disease; mass of any size permitted if positron emission tomography (PET) negative; regression to normal size on computed tomography (CT); spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy.
Time Frame: Up to 97 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 262 | 261
percentage of participants | 57.6 | 65.5

4. Secondary Outcome: Time-to-Next Treatment
Description: Time-to-next treatment was measured from the date of randomization to the start date of any anti-mantle cell lymphoma (anti-MCL) treatment subsequent to the study treatment.
Time Frame: Up to 97 months
Population: ITT analysis set included all randomized participants and classified according to the assigned treatment group, regardless of the actual treatment received. Here, N (number of participants analyzed) signifies number of participants that were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 262 | 261
months | 92.0 [71.5 to NA] — Here, 'NA' refers that the upper limit of 95% confidence interval was not estimable due to a small number of participants with events. | NA [NA to NA] — Here, 'NA' refers that the median and 95% confidence interval were not estimable due to a small number of participants with events.

5. Secondary Outcome: Percentage of Participants With Overall Response
Description: Percentage of participants with overall response was defined as the portion of participants who achieved CR or PR. Criteria for CR: disappearance of all evidence of disease; mass of any size permitted if PET negative; regression to normal size on CT; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy. Criteria for PR: greater than or equal to (>=) 50% decrease in sum of the diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions.
Time Frame: Up to 97 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 262 | 261
percentage of participants | 88.5 | 89.7

6. Secondary Outcome: Minimal Residual Disease (MRD)-Negative Response Rate
Description: Minimal residual disease negative rate was defined as the percentage of participants with a best overall response of CR with MRD-negative disease status (that is, <5 mantle cell lymphoma [MCL] cell per 10,000 leukocytes for detection using the MRD assay), as assessed by flow cytometry of a bone marrow and/or peripheral blood sample.
Time Frame: Up to 97 months
Population: ITT analysis set included all randomized participants and classified according to the assigned treatment group, regardless of the actual treatment received. CR participants with missing MRD data and participants who did not achieve a CR were considered nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 262 | 261
percentage of participants | 56.5 | 62.1

7. Secondary Outcome: Time to Worsening (TTW) in the Lymphoma (Lym) Subscale of the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) Questionnaire
Description: Time to worsening in the Lymphoma subscale of the FACT-Lym, defined as the interval from the date of randomization to the start date of worsening of participant symptoms. Worsening was defined by a 5-point decrease from baseline, death, or a missing assessment due to being "too ill", whichever occurred first. FACT-Lym Lymphoma subscale contains 15 questions, scores from 0 to 4 for each question (higher the worse). Lymphoma subscale score was the total of reverse scores, ranged 0 to 60. Higher scores indicated a better quality of life.
Time Frame: Up to 97 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 262 | 261
months | 22.2 [9.3 to 34.0] | 17.4 [8.3 to 27.6]

8. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DoR) was defined as the interval between the date of initial documentation of a response including PR and the date of first documented evidence of PD or death
Time Frame: Up to 97 months
Population: ITT analysis set included all randomized participants and classified according to the assigned treatment group, regardless of the actual treatment received. Participants who achieved a PR or better were included in the analysis of duration of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 232 | 234
months | 63.5 [47 to 76.9] | 81 [64.2 to NA] — Here, 'NA' refers that the upper limit of 95% confidence interval was not estimable due to a small number of participants with events.

9. Secondary Outcome: Duration of Complete Response (DoCR)
Description: Duration of complete response (DoCR) was defined as the interval between the date of initial documentation of a CR and the date of first documented evidence of PD or death whichever occurs first.
Time Frame: Up to 97 months
Population: ITT analysis set included all randomized participants and classified according to the assigned treatment group, regardless of the actual treatment received. Participants who achieved a CR or better were included in the analysis of duration of complete response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 151 | 171
months | 78.1 [65.6 to NA] — Here, 'NA' refers that the upper limit of 95% confidence interval were not estimable due to a small number of participants with events. | NA [81.7 to NA] — Here, 'NA' refers that the median and upper limit of 95% confidence interval were not estimable due to a small number of participants with events.

10. Secondary Outcome: Time to Response
Description: Time to response was defined as the interval between the date of randomization and the date of initial documentation of a response.
Time Frame: Up to 97 months
Population: ITT analysis set included all randomized participants and classified according to the assigned treatment group, regardless of the actual treatment received. Participants who achieved a PR or better were included in the analysis of time to response.
Measure: Median (Full Range); unit: months
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 232 | 234
months | 2.79 [1.9 to 11.2] | 2.79 [2.1 to 10.1]

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. Treatment-emergent adverse events were defined as adverse events with onset or worsening on or after date of first dose of study treatment up to and including 30 days after date of last dose of study medication, or the initiation of subsequent anticancer therapy, whichever is earlier.
Time Frame: Placebo + BR (Treatment A): From first dose of study treatment (Day 1) up to 100.1 months; Ibrutinib + BR (Treatment B): From first dose of study treatment (Day 1) up to 117.2 months
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug (ibrutinib or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 260 | 259
Participants | 257 | 259

12. Secondary Outcome: Oral Plasma Clearance (CL/F) of Ibrutinib
Description: CL/F was defined as apparent total systemic clearance of ibrutinib after extravascular administration. Cl/F of Ibrutinib was determined using population pharmacokinetics (PopPK modeling).
Time Frame: Pre-dose on Day 2 of Cycles 1, 2 and 3; and 1, 2 and 4 hours post-dose on Day 2 of Cycles 1 and 2
Population: Pharmacokinetic-evaluable population included participants who have received at least 1 dose of ibrutinib/placebo and had at least 1 pharmacokinetic sample obtained posttreatment.
Measure: Mean (Standard Error); unit: liter per hour (L/h)
Arm/Group | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 259
liter per hour (L/h) | 1123 (4.83)

13. Secondary Outcome: Oral Volume of Distribution at Steady State of Ibrutinib
Description: Oral volume of distribution at steady state of ibrutinib was determined using PopPK modeling.
Time Frame: Pre-dose on Day 2 of Cycles 1, 2 and 3; and 1, 2 and 4 hours post-dose on Day 2 of Cycles 1 and 2
Population: as for outcome 12
Measure: Mean (Standard Error); unit: liter
Arm/Group | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 259
liter | 7286 (7.87)

14. Secondary Outcome: Area Under the Concentration Curve of Ibrutinib During 24 Hours After Dosing at Steady State
Description: Area under the concentration curve of ibrutinib during 24 hours after dosing at steady state was determined using PopPK modeling.
Time Frame: Pre-dose on Day 2 of Cycles 1, 2 and 3; and 1, 2 and 4 hours post-dose on Day 2 of Cycles 1 and 2
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 259
nanogram*hour per milliliter (ng*h/mL) | 425 (267)

15. Secondary Outcome: Minimum Observed Plasma Concentration of Ibrutinib
Description: Minimum observed plasma concentration of ibrutinib was determined using PopPK modeling.
Time Frame: Pre-dose on Day 2 of Cycles 1, 2 and 3; and 1, 2 and 4 hours post-dose on Day 2 of Cycles 1 and 2
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 259
nanograms per milliliter (ng/mL) | 3.90 (2.64)

16. Secondary Outcome: Maximum Observed Plasma Concentration of Ibrutinib
Description: Maximum observed plasma concentration of ibrutinib was determined using PopPK modeling.
Time Frame: Pre-dose on Day 2 of Cycles 1, 2 and 3; and 1, 2 and 4 hours post-dose on Day 2 of Cycles 1 and 2
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
Number analyzed (Participants) | 259
ng/mL | 74.5 (48.3)

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization (Day -3) up to 121 months; SAEs and Non SAEs: Placebo + BR (Treatment A): From first dose of study treatment (Day 1) up to 100.1 months; Ibrutinib + BR (Treatment B): From first dose of study treatment (Day 1) up to 117.2 months
Description: All-cause mortality: All randomized participants. SAEs and Non SAEs: Safety analysis set included all randomized participants who received at least 1 dose of study drug (ibrutinib or placebo).
Arm/Group | Placebo + Bendamustine and Rituximab (BR) (Treatment A) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B)
All-Cause Mortality (participants affected / at risk) | 129/262 | 120/261
Serious Adverse Events (participants affected / at risk) | 157/260 | 201/259
Other Adverse Events (participants affected / at risk) | 255/260 | 256/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Bendamustine and Rituximab (BR) (Treatment A) (N=260) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B) (N=259)
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 | 16
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 3
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Splenic Infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 4 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 4 | 14
Atrial Flutter (Cardiac disorders) | 1 | 3
Atrioventricular Block (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 5
Cardiac Failure (Cardiac disorders) | 1 | 4
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 2 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 1 | 0
Mitral Valve Stenosis (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 6 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 2
Nodal Rhythm (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1
Silent Myocardial Infarction (Cardiac disorders) | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Sinus Node Dysfunction (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0
Odontogenic Cyst (Congenital, familial and genetic disorders) | 1 | 0
Hyperaldosteronism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Exophthalmos (Eye disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1
Ulcerative Keratitis (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 3
Acute Abdomen (Gastrointestinal disorders) | 0 | 1
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 8
Gastric Perforation (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 3
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 2 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4
Proctitis (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 5
Asthenia (General disorders) | 2 | 0
Chest Discomfort (General disorders) | 1 | 0
Chest Pain (General disorders) | 2 | 2
Chills (General disorders) | 1 | 1
Death (General disorders) | 0 | 3
Fatigue (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 4
Localised Oedema (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 3
Mucosal Inflammation (General disorders) | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 3
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 3
Pyrexia (General disorders) | 14 | 19
Sudden Death (General disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 2
Hypersensitivity (Immune system disorders) | 1 | 2
Serum Sickness (Immune system disorders) | 0 | 1
Abscess Intestinal (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 2 | 1
Arthritis Bacterial (Infections and infestations) | 1 | 0
Bacterial Sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 4 | 7
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 4
Campylobacter Gastroenteritis (Infections and infestations) | 1 | 1
Campylobacter Infection (Infections and infestations) | 0 | 1
Candida Sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 9
Clostridium Colitis (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 3
Covid-19 (Infections and infestations) | 0 | 3
Covid-19 Pneumonia (Infections and infestations) | 2 | 8
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus Colitis (Infections and infestations) | 0 | 1
Cytomegalovirus Infection (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 2 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Epididymitis (Infections and infestations) | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 2
Escherichia Bacteraemia (Infections and infestations) | 0 | 2
Escherichia Infection (Infections and infestations) | 0 | 1
Fungal Oesophagitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 4
Gastroenteritis Salmonella (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1
Hepatitis B Reactivation (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 3 | 3
Herpes Zoster Disseminated (Infections and infestations) | 0 | 1
Herpes Zoster Oticus (Infections and infestations) | 1 | 0
Histoplasmosis Disseminated (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 2 | 1
Listeriosis (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 0 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 5
Lung Abscess (Infections and infestations) | 0 | 1
Meningococcal Bacteraemia (Infections and infestations) | 0 | 1
Moraxella Infection (Infections and infestations) | 1 | 0
Nosocomial Infection (Infections and infestations) | 0 | 1
Oesophageal Candidiasis (Infections and infestations) | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 1
Oropharyngeal Candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Osteomyelitis Chronic (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 1
Parasitic Gastroenteritis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Periorbital Cellulitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumococcal Bacteraemia (Infections and infestations) | 1 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 35 | 58
Pneumonia Aspiration (Infections and infestations) | 0 | 1
Pneumonia Bacterial (Infections and infestations) | 2 | 1
Pneumonia Cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia Fungal (Infections and infestations) | 0 | 2
Pneumonia Pneumococcal (Infections and infestations) | 1 | 0
Pneumonia Pseudomonal (Infections and infestations) | 2 | 0
Pneumonia Viral (Infections and infestations) | 1 | 2
Postoperative Wound Infection (Infections and infestations) | 1 | 0
Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 1 | 0
Pseudomembranous Colitis (Infections and infestations) | 2 | 0
Pseudomonas Infection (Infections and infestations) | 0 | 1
Pulmonary Sepsis (Infections and infestations) | 1 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis Chronic (Infections and infestations) | 0 | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 5
Sepsis (Infections and infestations) | 6 | 10
Septic Shock (Infections and infestations) | 2 | 3
Sialoadenitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 4
Sinusitis Bacterial (Infections and infestations) | 0 | 1
Sinusitis Fungal (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 0 | 2
Soft Tissue Infection (Infections and infestations) | 2 | 2
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 2
Staphylococcal Infection (Infections and infestations) | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Streptococcal Bacteraemia (Infections and infestations) | 1 | 1
Suspected Covid-19 (Infections and infestations) | 0 | 1
Toxoplasmosis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 4
Urinary Tract Infection (Infections and infestations) | 2 | 7
Urosepsis (Infections and infestations) | 3 | 2
Vascular Device Infection (Infections and infestations) | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 2
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 2
Infusion Related Reaction (Injury, poisoning and procedural complications) | 4 | 2
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Stoma Complication (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 4 | 4
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 2
Blood Creatinine Increased (Investigations) | 2 | 0
Bronchoscopy (Investigations) | 0 | 1
Cytomegalovirus Test Positive (Investigations) | 1 | 1
Gastrointestinal Stoma Output Increased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 1
Platelet Count Decreased (Investigations) | 3 | 1
Scan Abnormal (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 5 | 4
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Finger Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaw Cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Appendix Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Benign Anorectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic Myelomonocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Langerhans' Cell Histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ocular Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin Squamous Cell Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 0 | 1
Brain Oedema (Nervous system disorders) | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 1
Central Nervous System Lesion (Nervous system disorders) | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0
Facial Paralysis (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 3
Lacunar Stroke (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Quadriplegia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 5
Thalamic Infarction (Nervous system disorders) | 1 | 0
Transient Global Amnesia (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 1
Vascular Encephalopathy (Nervous system disorders) | 0 | 1
Device End of Service (Product Issues) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 2 | 8
Calculus Urinary (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Renal Colic (Renal and urinary disorders) | 1 | 0
Renal Cyst Haemorrhage (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 3
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 2
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 2
Prostatic Obstruction (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypersensitivity Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Tonsillar Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Drug Reaction with Eosinophilia and Systemic Symptoms (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 5
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Coronary Artery Bypass (Surgical and medical procedures) | 1 | 0
Tracheostomy Closure (Surgical and medical procedures) | 1 | 0
Aortic Stenosis (Vascular disorders) | 1 | 0
Arterial Thrombosis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Giant Cell Arteritis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1
Hypertensive Urgency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 2
Peripheral Artery Aneurysm (Vascular disorders) | 0 | 1
Raynaud's Phenomenon (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Bendamustine and Rituximab (BR) (Treatment A) (N=260) | Ibrutinib + Bendamustine and Rituximab (BR) (Treatment B) (N=259)
Anaemia (Blood and lymphatic system disorders) | 60 | 83
Leukopenia (Blood and lymphatic system disorders) | 14 | 27
Lymphopenia (Blood and lymphatic system disorders) | 14 | 18
Neutropenia (Blood and lymphatic system disorders) | 104 | 109
Thrombocytopenia (Blood and lymphatic system disorders) | 43 | 62
Atrial Fibrillation (Cardiac disorders) | 14 | 32
Palpitations (Cardiac disorders) | 13 | 9
Vertigo (Ear and labyrinth disorders) | 13 | 11
Cataract (Eye disorders) | 17 | 21
Dry Eye (Eye disorders) | 5 | 16
Vision Blurred (Eye disorders) | 10 | 14
Abdominal Pain (Gastrointestinal disorders) | 29 | 25
Abdominal Pain Upper (Gastrointestinal disorders) | 10 | 19
Constipation (Gastrointestinal disorders) | 66 | 52
Diarrhoea (Gastrointestinal disorders) | 96 | 119
Dry Mouth (Gastrointestinal disorders) | 6 | 18
Dyspepsia (Gastrointestinal disorders) | 21 | 21
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 16 | 18
Nausea (Gastrointestinal disorders) | 107 | 109
Stomatitis (Gastrointestinal disorders) | 6 | 23
Vomiting (Gastrointestinal disorders) | 48 | 56
Asthenia (General disorders) | 25 | 30
Chest Pain (General disorders) | 12 | 14
Chills (General disorders) | 39 | 17
Fatigue (General disorders) | 77 | 79
Influenza Like Illness (General disorders) | 13 | 14
Malaise (General disorders) | 14 | 12
Mucosal Inflammation (General disorders) | 15 | 14
Oedema Peripheral (General disorders) | 42 | 50
Pyrexia (General disorders) | 76 | 88
Hypogammaglobulinaemia (Immune system disorders) | 14 | 9
Bronchitis (Infections and infestations) | 36 | 33
Cellulitis (Infections and infestations) | 4 | 15
Conjunctivitis (Infections and infestations) | 6 | 26
Covid-19 (Infections and infestations) | 3 | 17
Herpes Zoster (Infections and infestations) | 27 | 15
Influenza (Infections and infestations) | 16 | 9
Lower Respiratory Tract Infection (Infections and infestations) | 9 | 13
Nasopharyngitis (Infections and infestations) | 28 | 25
Oral Candidiasis (Infections and infestations) | 7 | 19
Pneumonia (Infections and infestations) | 39 | 53
Rhinitis (Infections and infestations) | 13 | 10
Sinusitis (Infections and infestations) | 34 | 25
Skin Infection (Infections and infestations) | 5 | 18
Upper Respiratory Tract Infection (Infections and infestations) | 69 | 70
Urinary Tract Infection (Infections and infestations) | 32 | 36
Contusion (Injury, poisoning and procedural complications) | 12 | 23
Fall (Injury, poisoning and procedural complications) | 13 | 16
Infusion Related Reaction (Injury, poisoning and procedural complications) | 26 | 19
Alanine Aminotransferase Increased (Investigations) | 12 | 23
Aspartate Aminotransferase Increased (Investigations) | 14 | 24
Blood Creatinine Increased (Investigations) | 22 | 23
Lymphocyte Count Decreased (Investigations) | 26 | 32
Neutrophil Count Decreased (Investigations) | 43 | 39
Platelet Count Decreased (Investigations) | 28 | 41
Weight Decreased (Investigations) | 20 | 26
White Blood Cell Count Decreased (Investigations) | 34 | 30
Decreased Appetite (Metabolism and nutrition disorders) | 36 | 54
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 15
Hyperuricaemia (Metabolism and nutrition disorders) | 20 | 24
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 30 | 39
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 46
Back Pain (Musculoskeletal and connective tissue disorders) | 38 | 36
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 13 | 21
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 5 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 30 | 33
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 24 | 18
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 12
Dizziness (Nervous system disorders) | 19 | 22
Headache (Nervous system disorders) | 40 | 33
Paraesthesia (Nervous system disorders) | 13 | 13
Anxiety (Psychiatric disorders) | 17 | 14
Depression (Psychiatric disorders) | 12 | 16
Insomnia (Psychiatric disorders) | 28 | 29
Haematuria (Renal and urinary disorders) | 7 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 85 | 78
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45 | 27
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 31
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 7
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 24 | 23
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 16
Dry Skin (Skin and subcutaneous tissue disorders) | 11 | 21
Erythema (Skin and subcutaneous tissue disorders) | 12 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 56 | 47
Rash (Skin and subcutaneous tissue disorders) | 57 | 95
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 10 | 22
Skin Lesion (Skin and subcutaneous tissue disorders) | 11 | 16
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 16
Haematoma (Vascular disorders) | 3 | 20
Hypertension (Vascular disorders) | 29 | 37
Hypotension (Vascular disorders) | 16 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT01776840/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT01776840/SAP_001.pdf